CLINICAL TRIAL: NCT05401175
Title: Stored Hematopoietic Stem Cell-containing Autologous Blood Transfusion Therapy for Bone Marrow Protection in Patients With Cervical Cancer Treated With Concurrent Chemoradiotherapy
Brief Title: Hematopoietic Stem Cell-containing Autologous Blood Transfusion for Bone Marrow Protection in Patients With Cervical Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chongqing University Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQGOG0107
Record Dates: First submitted 2022-05-29; First posted 2022-06-02 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2022-09

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; concurrent chemoradiotherapy; blood stem cells; autologous blood transfusion
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Blood Transfusion, Autologous

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous blood transfusion support therapy group (Experimental): Bone aspiration and bone marrow examination before concurrent chemoradiotherapy.Peripheral blood stem cells were mobilized, frozen and stored before treatment. Resuscitate and reinfusion autologous peripheral blood 24 hours after completion of concurrent chemoradiotherapy.
  Interventions: Other: Autologous blood transfusion with haematopoietic stem cells
- Conventional treatment group (No Intervention): Bone aspiration and bone marrow examination before concurrent chemoradiotherapy.Undergo standard radiotherapy for cervical cancer.

INTERVENTIONS:
Other: Autologous blood transfusion with haematopoietic stem cells — Transfusion of autologous blood containing haematopoietic stem cells for haematopoietic reconstruction after chemoradiotherapy.Blood tests were performed weekly, if the patient's neutrophils were less than 1.0 × 109 / L during chemoradiotherapy, G-CSF was given as a remedial treatment. If fever occurs, antibiotics were given promptly.Monitor peripheral blood after transfusion. If peripheral blood leukocyte count does not reach 1.0 x 109/L, administer G-CSF 150 μg subcutaneously daily until peripheral blood leukocyte count reaches 1.0 x 109/L.Patients were tested monthly for peripheral blood cells for 6 months after the end of treatment.
  Arms: Autologous blood transfusion support therapy group

SUMMARY:
The aim of this project is to promote the reconstruction of haematopoietic function after chemoradiotherapy for cervical cancer with the innovative use of autologous haematopoietic containing stem cell blood transfusion support.To explore the effect of stored hemopoietic stem cell support therapy on bone marrow protection after concurrent chemoradiotherapy, in order to promote its clinical application.

DETAILED DESCRIPTION:
Study design:In this prospective, single-center,non-randomised controlled study, patients with cervical cancer are divided into two groups. Patients in the autologous blood transfusion support therapy group will receive autologous blood transfusion containing haematopoietic stem cells after completion of concurrent chemoradiotherapy, whereas the conventional treatment group receive concurrent chemoradiotherapy only. Frozen stored autologous peripheral blood transfusion 1 day after completion of chemoradiotherapy.Monitor peripheral blood after transfusion. If peripheral blood leukocyte count does not reach 1.0 x 109/L, administer G-CSF 150 μg subcutaneously daily until peripheral blood leukocyte count reaches 1.0 x 109/L.

Case selection: Patients with primary cervical cancer,squamous, adenocarcinoma or adenosquamous carcinoma cell carcinoma confirmed by histopathology, and three-week regimen of paclitaxel and platinum chemotherapy with concurrent radiotherapy.

Primary end point: 1)incidence and duration of grade 3/4 neutropenia in patients;2)hematopoietic reconstitution time in patients. Secondary endpoints: 1)the rate of postponement of the course of radiotherapy, reduction in chemotherapy dose and postponement of the course of chemotherapy;2) Incidence of febrile neutropenia (FN);3)Safety of hematopoietic stem cell reinfusion therapy (adverse events).

Safety assessment: laboratory safety testing, including platelet count,white blood cell and hemoglobin. Evaluation of adverse events: infection, neutropenic fever, hypocalcemia,anemia and thrombocytopenia,bone pain, etc.

ELIGIBILITY:
Inclusion Criteria:

1）18-60 years old; 2)there are radiotherapy and chemotherapy indicators for cervical cancer;3)pathological diagnosis of squamous, adenocarcinoma or adenosquamous carcinoma;4)the Eastern Cooperative Oncology Group (ECOG) performance status score≤1; 5)the expected survival time was more than 3 months; 6)pre-menopausal women (post-menopausal women must have been postmenopausal for at least 12 months to be considered infertile), and the serum pregnancy test results are negative;7)all patients must agree to take effective contraceptive measures during the study period and within 6 months after stopping treatment;8)the subjects voluntarily participate in this clinical trial sign an informed consent form and are able to complete the study procedures and follow-up examinations.

Exclusion Criteria:

1) clinical diagnosis of bone marrow disease;2) imaging or pathological diagnosis of central nervous system or soft meningeal or bone or bone marrow metastases;3)patient has severe cardiac insufficiency;4)previous history of allogeneic stem cell transplantation or organ transplantation;5)patients with active bleeding and autoimmune thrombocytopenic purpura;6)patients with radiochemotherapy contraindications;7)positive for human immunodeficiency virus (HIV);8)acute or chronic active hepatitis B or hepatitis C infection;9)History of gastrointestinal perforation and/or fistula, clinical signs or symptoms of intestinal obstruction and/or gastrointestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), inflammatory bowel disease or extensive bowel resection (partial colectomy or extensive small bowel resection complicated by chronic diarrhoea), Crohn's disease, ulcerative colitis or chronic diarrhoea within the previous 6 months;10)evidence of an intra-abdominal pneumoperitoneum that cannot be explained by puncture or recent surgical intervention.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-13 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade 3-4 neutropenia | 6 months
  Incidence of Grade 3-4 neutropenia
Time to reconstruct haematopoietic function | 6 months
  Time to reconstruct haematopoietic function

SECONDARY OUTCOMES:
the rate of postponement of the course of chemoradiotherapy | 3 months
  the rate of postponement of the course of chemoradiotherapy
reduction in chemotherapy dose | 3 months
  reduction in chemotherapy dose
Incidence of febrile neutropenia (FN) | 3 months
  Incidence of febrile neutropenia (FN)
Incidence of hematopoietic stem cell reinfusion treatment Adverse Events [Safety and Tolerability]) | 1 months
  Incidence of hematopoietic stem cell reinfusion treatment Adverse Events [Safety and Tolerability])

CONTACTS AND LOCATIONS:
Overall Officials: Dongling Zou, M.D., Principal Investigator — Chongqing University Cancer Hospital
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bhargava A, Mishra DK, Jain SK, Srivastava RK, Lohiya NK, Mishra PK. Comparative assessment of lipid based nano-carrier systems for dendritic cell based targeting of tumor re-initiating cells in gynecological cancers. Mol Immunol. 2016 Nov;79:98-112. doi: 10.1016/j.molimm.2016.10.003. Epub 2016 Oct 17. PMID 27764711
- [Background] Huang BH, Li J, Zou WY, Liu JR, Gu JL, Li XZ, Chen ML, Kuang LF. [Efficacy and safety of autologous hematopoietic stem cell transplantation in elderly multiple myeloma patients: a single center retrospective study]. Zhonghua Xue Ye Xue Za Zhi. 2022 Feb 14;43(2):141-145. doi: 10.3760/cma.j.issn.0253-2727.2022.02.009. Chinese. PMID 35381675
- [Background] Fares S, Hadri H, Rachid M, Moutiqui T, Oukkache B, Quessar A. [Multiple myeloma and autologous haematopoietic stem-cell transplantation without cryopreservation: experiences of the Clinical Hematology Department of Casablanca, Morocco]. Pan Afr Med J. 2021 Jun 4;39:105. doi: 10.11604/pamj.2021.39.105.18994. eCollection 2021. French. PMID 34512841
- [Background] Corbeau A, Kuipers SC, de Boer SM, Horeweg N, Hoogeman MS, Godart J, Nout RA. Correlations between bone marrow radiation dose and hematologic toxicity in locally advanced cervical cancer patients receiving chemoradiation with cisplatin: a systematic review. Radiother Oncol. 2021 Nov;164:128-137. doi: 10.1016/j.radonc.2021.09.009. Epub 2021 Sep 21. PMID 34560187